CLINICAL TRIAL: NCT02157168
Title: Connecting Healthy Women: Examining the Effect of an Intervention From the Effect of Being Reachable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IHS-1306-04356
Record Dates: First submitted 2014-05-29; First posted 2014-06-05 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2017-03

CONDITIONS: Contraception; Sexually Transmitted Infections; Cervical Cancer
Keywords: Affordable Care Act; Medically underserved minorities; Community health workers; Health disparities among Mexican origin
MeSH Terms: conditions — Sexually Transmitted Diseases; Uterine Cervical Neoplasms | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Each month all newly enrolled female health plan members will have an equal chance of being randomly picked by the health plan (according to a randomization scheme provided by the study team) to be invited to contact and work with a Community health worker. Those not invited will constitute the usual care control group.
- Intervention Group (Other): Each month all newly enrolled female health plan members will have an equal chance of being randomly picked by the health plan (according to a randomization scheme provided by the study team) to be invited to contact and work with a Community health worker in the intervention group.
  The intervention group will be made up of two sub groups. The group of individuals who accept the invitation to participate (IG1) in the intervention and receive it, and those randomized to the intervention group but who reject the opportunity to participate (IG2).
  Interventions: Behavioral: Community health worker

INTERVENTIONS:
Behavioral: Community health worker — Community health workers (CHWs) in Hispanic communities, often referred to as "promotoras," are members of the community who use "resource sharing, partnership development, education, outreach, health promotion, and disease prevention strategies to improve the health" of their communities.
  IG1: The intervention itself consists of a 45-minute one-on-one presentation and tailored planning session delivered by a CHW in a community setting of the new member's choosing. Presentations (in English or Spanish) will be delivered using a tablet computer or a hand held flipchart. Two booster telephone interactions will be performed at 2 and 4 months. At month 6, the participant will receive a call from the telephone interviewer to administer the informed patient choice survey.
  Other Names: Promotoras
  Arms: Intervention Group

SUMMARY:
The investigators propose to test a community-developed and targeted intervention that employs community health workers (CHWs) as aides to newly Medicaid-insured women. These women face the challenges of engaging with their healthcare and health and of making highly personal and socioculturally embedded decisions about reproductive health-related preventive services (e.g., contraception, STI and cancer screening).

DETAILED DESCRIPTION:
All newly enrolled women in one of Arizona's state-wide Medicaid health plans (University Family Care) who are ambulatory and community-dwelling, and between the ages of 18-39, will be identified by the health plan on a monthly basis as eligible for this study. For at least the first month, these new health plan members will be randomized 2 to 1 (intervention to usual care control). Each month the health plan will provide the study team with the number of new members. A study team member will then provide the health plan with a list of numbers (1's and 0's) generated using the biased coin design to apply to those new members. To avoid bias, health plan staff will not be aware of members study arm.

All new health plan enrollees (as per current standard health plan practice) receive a series of welcome communications (by mail and electronically) from the health plan shortly after enrollment. These are designed to apprise new members of health plan policies and procedures related to covered benefits, facilitate the selection of a primary care provider, and provide general preventive health resources and information. This is followed by a second mailing at 3-months post enrollment, as well as a nurse follow-up call. The latter is designed to answer questions about covered services, finding a primary care provider, and/or otherwise provide support. Both intervention and control group member will receive identical communications from the health plan up to this point. Potential participants will be contacted by the health plan's call center. A brief verbal overview of the intervention including time requirement and content to be covered will be provided. The potential participants who have been randomly assigned to the intervention group will then be offered the opportunity to set up an individual confidential appointment with a community health worker (CHW) at her earliest convenience.

The call center will provide the research office a list of interested participants and their contact information. Once that list is received by the research office, a CHW will be assigned to each potential participant. The assigned CHW will call to introduce herself, to answer lingering questions about the intervention and proposed encounter and to confirm the participant's acceptance into the intervention. At that time, the CHW will confirm language and location preference, date/ time of proposed meeting, and the contact information for the research office for any questions. The CHW will meet with the subject and complete the informed consent process. Also, the baseline informed patient choice survey will be performed using a touch tablet device (to ascertain baseline knowledge, patient preferences, informed decision making, and health literacy). The CHW will tailor the individual education session to meet the unique needs of the participant (e.g., an individual who discloses a history of surgical sterilization will not receive information about contraception). The 45-minute intervention will be delivered as described above. The patient will be asked to personally assess her needs with regard to reproductive health-related issues. The CHW will work with the participant to develop a personalized plan to access the relevant targeted preventive services. This may involve assistance with contacting the Health Plan and assistance with identifying or making an appointment with a primary care provider. At the conclusion of the intervention, the patient will be encouraged to reach out to the CHW by telephone or electronically if she has any subsequent questions or concerns, and appointments for the two booster telephone calls will be scheduled. Finally, in consideration for her time and participation, the participant will be provided with a $40 gift card.

Booster telephone support calls will occur at 2 and 4 months post intervention. A telephone call guide will be used to reinforce and clarify key concepts from the initial intervention encounter as well as to help clients formulate relevant questions related to specific women's preventive services and other health concerns in anticipation of their next primary care provider (PCP) visit. Participants will also be queried specifically about any issues related to interactions with the health plan and/or contacting her primary care provider. The patient will be assisted with connecting to the health plan or her PCP's office for those issues that cannot be easily addressed by the CHW. Whenever possible, every effort will be made by the CHW to connect the patient to the appropriate outreach staff at that PCP's office (if such staff is available). Again the availability of the CHW by telephone or electronically for interval questions will be emphasized. At month 6, the participant will receive a call from the telephone interviewer to administer the 6-month informed patient choice survey identical to the survey that was completed at baseline. A $40 gift card incentive will be offered to complete this survey.

The call center will administer a similar 6-month survey by phone to a sample of the group randomized to invitation, but who did not accept the invitation (IG2) and the group not invited (CG). A $30 gift card incentive will be offered to complete this survey.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 39
* Women newly enrolled in one of the state-wide Medicaid health plans (University Family Care)
* Women who are ambulatory
* Women who are community-dwelling

Exclusion Criteria:

* Women not between the ages of 18 and 39
* Women not newly enrolled in one of the state wide Medicaid health plans (University Family Care)
* Women who are not ambulatory
* Women who are not community dwelling

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2267 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franciso AR Garcia, MD, MPH, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each month all newly enrolled female health plan members were randomly picked by the health plan (according to a randomization scheme provided by the study team) to be invited to work with a community health worker (CHW). Those not invited constituted the usual care control group. Recruitment began March 2015 and ended May 2016.
Groups:
- Control Group (CG): Each month all newly enrolled female health plan members had an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker. Those not invited constituted the usual care control group.
- Intervention Group (IG1): Each month all newly enrolled female health plan members had an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker in the intervention group.
  The intervention group was made up of two sub groups. The IG1 group is made up of those individuals who accept the invitation to participate in the intervention and receive it.
- Intervention Group (IG2): Each month all newly enrolled female health plan members had an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker in the intervention group.
  The intervention group was made up of two sub groups. The IG2 group is comprised of those randomized to the intervention group but who reject the opportunity to participate.
Period: Overall Study
Arm/Group | Control Group (CG) | Intervention Group (IG1) | Intervention Group (IG2)
Started | 746 | 159 | 1362
Completed | 746 | 159 | 1362
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (CG) | Intervention Group (IG1) | Intervention Group (IG2) | Total
Number analyzed (Participants) | 746 | 159 | 1362 | 2267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 746 | 159 | 1362 | 2267
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (6.0) | 28.5 (5.9) | 27.0 (6.1) | 27.2 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 746 | 159 | 1362 | 2267
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 218 | 70 | 431 | 719
  Not Hispanic or Latino | 423 | 62 | 736 | 1221
  Unknown or Not Reported | 105 | 27 | 195 | 327
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 41 | 1 | 60 | 102
  Asian | 15 | 0 | 23 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 61 | 9 | 123 | 193
  White | 523 | 122 | 961 | 1606
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 105 | 27 | 195 | 327
Region of Enrollment [Number; unit: participants]
  United States | 746 | 159 | 1362 | 2267

OUTCOME MEASURES:

1. Primary Outcome: Identify and Utilization of Primary Care Provider (PCP)
Description: The number and percentage of new members who had at least one visit with a primary care provider during their first 6 months of enrollment.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (CG) | Intervention Group (IG1) | Intervention Group (IG2)
Number analyzed (Participants) | 746 | 159 | 1362
Participants | 426 | 114 | 771
Statistical Analysis 1: Comparison: Control Group (CG) vs Intervention Group (IG1) vs Intervention Group (IG2); CG and IG (IG1+IG2); Test type: Superiority; p = 0.624, Chi-squared — This comparison reflects intent to treat and is the main comparison in the study
Statistical Analysis 2: Comparison: Control Group (CG) vs Intervention Group (IG1); Test type: Superiority; p = 0.001, Chi-squared — This comparison could be considered to be a per protocol analysis. Note, however, that the IG1 group was self-selected

2. Secondary Outcome: The Impact of the Intervention on the Utilization of Women's Preventive Services and Other Preventive Services
Description: The number and percentage of new members who had at least one preventive visit (i.e., well woman visit, cervical cancer screening, sexually transmitted infection (STI) screening, STI counseling, contraception counseling or immunizations) during their first 6 months of enrollment.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (CG) | Intervention Group (IG1) | Intervention Group (IG2)
Number analyzed (Participants) | 746 | 159 | 1362
Participants | 189 | 52 | 366
Statistical Analysis 1: Comparison: Control Group (CG) vs Intervention Group (IG1) vs Intervention Group (IG2); CG and IG (IG1+IG2); Test type: Superiority; p = 0.278, Chi-squared — This comparison reflects intent to treat and compares the two randomized groups CG and IG (IG1+IG2)
Statistical Analysis 2: Comparison: Control Group (CG) vs Intervention Group (IG1); Test type: Superiority; p = 0.056, Chi-squared — This comparison could be considered to be a per protocol analysis. Note, however, that the IG1 group was self-selected

3. Secondary Outcome: The Impact of the Intervention on the Utilization of Avoidable Emergency Department (ED) Visits
Description: The number and percentage of new members who had avoidable emergency department (ED) visits during their first 6 months of enrollment.
Time Frame: 6 months
Population: Members who had an ED visit during the first 6 months of their enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (CG) | Intervention Group (IG1) | Intervention Group (IG2)
Number analyzed (Participants) | 467 | 88 | 767
Participants | 135 | 23 | 220
Statistical Analysis 1: Comparison: Control Group (CG) vs Intervention Group (IG1) vs Intervention Group (IG2); CG and IG (IG1+IG2); Test type: Superiority; p = 0.889, Chi-squared — This comparison reflects intent to treat and compares the two randomized groups CG and IG (IG1+IG2)
Statistical Analysis 2: Comparison: Control Group (CG) vs Intervention Group (IG1); Test type: Superiority; p = 0.691, Chi-squared — This comparison could be considered to be a per protocol analysis. Note, however, that the IG1 group was self-selected

4. Secondary Outcome: The Impact of the Intervention on Preventable Hospital Stays
Description: The number and percentage of new members who had avoidable hospitalizations during their first 6 months of enrollment.
Time Frame: 6 months
Population: Members who had a hospital visit during the first 6 months of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (CG) | Intervention Group (IG1) | Intervention Group (IG2)
Number analyzed (Participants) | 76 | 24 | 167
Participants | 13 | 4 | 25
Statistical Analysis 1: Comparison: Control Group (CG) vs Intervention Group (IG1) vs Intervention Group (IG2); CG and IG (IG1+IG2); Test type: Superiority; p = 0.741, Chi-squared — This comparison reflects intent to treat and compares the two randomized groups CG and IG (IG1+IG2)
Statistical Analysis 2: Comparison: Control Group (CG) vs Intervention Group (IG1); Test type: Superiority; p = 0.966, Chi-squared — This comparison could be considered to be a per protocol analysis. Note, however, that the IG1 group was self-selected

5. Other Pre Specified Outcome: Informed Decision Making Regarding the Healthcare System and Their Health
Description: The short form of the Patient Activation Measure (PAM), a measure of patient engagement in their healthcare. PAM levels of engagement with Level 4 being the highest level.
Time Frame: Baseline and 6 months
Population: IG1 group members that completed the baseline and 6-month survey and CG and IG2 group members that complete the 6-month survey.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Intervention Group (IG1): Each month all newly enrolled female health plan members had an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker in the intervention group.
  IG1 at Baseline: The intervention group was made up of two sub groups. The IG1 group is made up of those individuals who accept the invitation to participate in the intervention and receive it.
- 6-Month Follow-up: Intervention Group (IG1): Each month all newly enrolled female health plan members had an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker in the intervention group.
  IG1 at 6-Month Follow-up: The intervention group was made up of two sub groups. The IG1 group is made up of those individuals who accept the invitation to participate in the intervention and receive it.
- 6-Month Follow-up: Control Group (CG)&Intervention Group (IG2): Each month all newly enrolled female health plan members had an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker.
  CG and IG2 at 6-Month Follow-up: Those not invited constituted the usual care control group (CG). The intervention group was made up of two sub groups. The IG2 group is comprised of those randomized to the intervention group but who reject the opportunity to participate.
Arm/Group | Baseline: Intervention Group (IG1) | 6-Month Follow-up: Intervention Group (IG1) | 6-Month Follow-up: Control Group (CG)&Intervention Group (IG2)
Number analyzed (Participants) | 101 | 101 | 111
Participants
  1: Believes active role important | 8 | 1 | 2
  2: Confidence and knowledge to take action | 7 | 6 | 8
  3: Taking action | 38 | 41 | 36
  4: Staying the course under stress | 48 | 53 | 65
Statistical Analysis 1: Comparison: Baseline: Intervention Group (IG1) vs 6-Month Follow-up: Intervention Group (IG1); Test type: Superiority; p = .117, Chi-squared — This comparison captures the change over the intervention period
Statistical Analysis 2: Comparison: 6-Month Follow-up: Intervention Group (IG1) vs 6-Month Follow-up: Control Group (CG)&Intervention Group (IG2); Test type: Superiority; p = .638, Chi-squared — This comparison is an indication of whether the change seen between baseline and 6 months in the IG1 was due to the intervention or simply due to 6 months' enrollment

ADVERSE EVENTS:
Time Frame: Reported Adverse Events started the first day of randomization (March 2015) into the study and concluded on the last day of data collection (December 2016).
Groups:
- Control Group (CG): Each month all newly enrolled female health plan members will have an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker. Those not invited will constitute the usual care control group.
- Intervention Group (IG1): Each month all newly enrolled female health plan members will have an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker in the intervention group.
  The intervention group will be made up of two sub groups. The IG1 group is made up of those individuals who accept the invitation to participate in the intervention and receive it.
- Intervention Group (IG2): Each month all newly enrolled female health plan members will have an equal chance of being randomly picked by the health plan to be invited to contact and work with a community health worker in the intervention group.
  The intervention group will be made up of two sub groups. The IG2 group is comprised of those randomized to the intervention group but who reject the opportunity to participate.
Arm/Group | Control Group (CG) | Intervention Group (IG1) | Intervention Group (IG2)
Serious Adverse Events (participants affected / at risk) | 0/746 | 0/159 | 0/1362
Other Adverse Events (participants affected / at risk) | 0/746 | 0/159 | 0/1362

LIMITATIONS AND CAVEATS:
The health plan was unable to contact the majority of the population to make the offer of CHW services, and the young, generally healthy population made impacts on avoidable ED visits and hospitalizations difficult to detect within a 6 month period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT02157168/Prot_000.pdf